CLINICAL TRIAL: NCT04189653
Title: Clinical Outcomes After Implementation of Continuous Vital Sign Monitoring on the General Ward.
Acronym: COCOMO
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-4330
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2019-11

CONDITIONS: Clinical Deterioration
Keywords: Early Warning Scores; Continuous Vital Sign Monitoring; Escalation of Care; ICU-Transfer; Deterioration prevention
MeSH Terms: conditions — Clinical Deterioration | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Ward Inpatients 2017-2018: ALL General Ward Inpatients on our Gastro-Enterology Surgery ward and Internal Medicine ward in the period august 1st 2017-august 31st 2018.
- General Ward Inpatients 2018-2019: ALL General Ward Inpatients on our Gastro-Enterology Surgery ward and Internal Medicine ward in the period august 1st 2018-august 31st 2019.
  Interventions: Other: Continuous Monitoring

INTERVENTIONS:
Other: Continuous Monitoring — Wireless continuous vital sign monitoring (HR, RR, SBP/DBP, SAT)
  Groups: General Ward Inpatients 2018-2019

SUMMARY:
In 2018, continuous monitoring (CM) of 5 vital signs with a wearable device, including automated MEWS calculation within the EMR were introduced on the surgical and internal medicine ward of our hospital. Rather than taking the measurements manually, this enabled the nurses to periodically validate the continuously derived vital signs at the protocolled moments, and simultaneously get an automatically calculated MEWS reading,. Moreover, continuous vital sign monitoring provides single channel alarms and trends of the vital signs in between the regular measurement moments. Compared to periodic manual measurements and registration in the EMR, the continuous vital sign monitoring and automated MEWS calculations in the EMR may result in better identification of clinical deterioration, and may improve clinical outcome.

The primary objective of this study is to evaluate changes in total hospital and ward stay, "Total Events" during admission (rapid response team (RRT) calls and unexpected intensive care unit (uICU) admissions and deaths) after implementation of CM on the regular surgical and internal medicine wards. Secondary objective is to evaluate changes in MEWS scores at the moment of the uICU admissions, length of hospital, ward and ICU stay and the proportion of RRT calls that results in a ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Admission on Inclusion ward.

Exclusion Criteria:

* Opt out of file study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult general ward patients of the GE-surgery and Internal Medicine wards of a Dutch tertiary academic hospital.
Sampling Method: Probability Sample
Enrollment: 3896 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Unexpected Intensive Care Unit Admissions | During ward admission, from moment of arival on ward till discharge or transfer, average of 4 days.
  Unexpected Intensive Care Unit Admissions
Rapid Response Team Activations | During ward admission, from moment of arival on ward till discharge or transfer, average of 4 days.
  Rapid Response Team Activations

SECONDARY OUTCOMES:
Length of Stay | During ward, ICU and hospital admission, till discharge, transfer to other hospital or death. Average of 5 days.
  Length of stay on the ward, ICU and Hospital stay as whole

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided